CLINICAL TRIAL: NCT05503654
Title: Effect of Nutrition Education Delivered Through Gada System Leaders On Nutrition And Health Status Of Infants And Young Child In East Wollega Zone, Oromiya Regional State, Western Ethiopia: A Cluster Randomized Controlled Trial
Brief Title: To Evaluate the Effect of Nutrition Education on Infants and Young Children's Nutritional and Health Status in East Wollaga Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Tadele Amente, Principal Investigator, Jimma University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10082022
Record Dates: First submitted 2022-08-11; First posted 2022-08-17 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Education on Feeding and Health Status
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A two-arm parallel cluster randomized community trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Intervention Arm is an arm in which nutrition education will be given to caregivers of infants and young children less than two years aged using the Health Belief Model and Theory of Planned Behavior.
  Interventions: Behavioral: Nutrition education
- Control group (No Intervention): Control Arm is an arm to which the intervention will not be implemented.

INTERVENTIONS:
Behavioral: Nutrition education — Those interventional groups will take nutrition education by Gada System leaders for 6 consecutive months
  Arms: intervention group

SUMMARY:
Child undernutrition is the principal cause of child morbidity and mortality worldwide. It manifests in different forms including stunting, wasting, underweight, and micronutrient deficiencies. Globally, in 2020 it is estimated that 149.2 million of children under 5 years of age were affected by stunting, 45.4 million were suffering from wasting and 38.9 million were overweight. The actual figures, particularly for stunting and wasting, are expected to be higher due to the effects of the COVID-19 pandemic.

In spite of WHO and UNICEF recommendations on infants and young child feeding globally, 31% of children 6-8 months have not yet begun to eat complementary foods, and 81% of children aged 6-23 months are not fed the minimum acceptable diet (MAD). Inappropriate infant and young child feeding are a key causal factor in the development of malnutrition that increases the risk of undernutrition, illness, and mortality in infants and young children under five years, even more, severe in those less than 2 years of age because over two third of malnutrition is associated with inappropriate feeding practices during the first year of life.

The first two years of life provide a critical window of opportunity for ensuring appropriate growth and development of children from generation to generation through optimal feeding. Therefore, the aim of this study is to evaluate the effectiveness of nutrition education delivered through Gada System leaders on nutrition and the health status of infants and young children.

A Cluster randomized controlled trial design with two parallel arms among caregivers of infants and young children aged less than two years will be employed in East Wallaga Zone, Western Oromia, Ethiopia from October 01/2021 to November 30/2023. The intervention duration will be 6 months. A total of 566 mother-child dyads will be selected from eighteen kebeles via multi-stage cluster sampling methods. Pre-tested, structured, and interviewer-administered questionnaire will be used to collect data by trained data collectors. The collected data will be cleaned and checked for completeness, then enter into EpiData version 4.1 software to minimize error, then export to SPSS version 25 software for further analysis. Descriptive statistics and advanced analytics models including GEE and LMM will be used by checking the necessary assumption for each model.

The output of the study findings could be useful for health and nutrition policymakers and other concerned bodies in decision making and to design effective intervention strategies to improve feeding practices thus mitigating child malnutrition and improving their health and growth. The total budget required to conduct the study will be 7,420 US dollar

ELIGIBILITY:
Inclusion Criteria:

* All infants and young children aged 6-17 months at the time of the baseline survey
* Residents in the sampled kebeles

Exclusion Criteria:

* Mothers who are ill and unable to communicate
* Infants and young children with birth defects, impaired feeding, twin and ill at the time of baseline survey.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Core indicators of CF.Practices (i.e.. Minimum dietary diversity, minimum meal frequency, and minimum acceptable diet) | Baseline survey
  The developed questionnaire will be categorized according to World Health Organization and United Nations International Children Emergency Fund recommending guideline to assess the outcome variables.
  1. Minimum dietary diversity: if the child is between 6-23 months of age consumed equal or greater than 5 food groups from 8 food groups during the previous day
  2. Minimum meal frequency: If the children between 6-23 months of age consumed solid, semi-solid, or soft foods (but also including milk feeds for non-breastfed children) at least the minimum number of times(i.e.. 3 for breastfeeding, and 4 for non-breastfeed) during the previous day
  3. Minimum acceptable diet: If the children between 6-23 months of age consumed a minimum acceptable diet (i.e. fulfill minimum dietary diversity and minimum meal frequency for breast feed, and non-breastfeed) during the previous day.
Minimum Dietary diversity score | 6 months of intervention
  From the already developed questionnaire will be used to measure the change of dietary diversity between the baseline assessment and end-line assessment between and within the study groups after intervention according to World Health Organization recommendation guideline to measure the outcome variable.

SECONDARY OUTCOMES:
Child growth | 6 months of intervention
  Change in length (cm) and weight(kg) after intervention based on anthropometric measurement. Our target here is to assess the children between 6 and 23 months old; baseline and end-line anthropometric data will be collected from all participants. Child physical growth will be considered an outcome measure, measured by length gain (i.e., end-line minus baseline length in centimeters), and weight gain (i.e, end-line minus baseline weight in kilograms) separately, and reported under one objective separately. The aim is not to create a composite variable like BMI.
Morbidity status | 6 months of intervention
  The questionnaire adopted from the Ethiopian Demographic and Health Survey report of 2016 will be used to assess the outcome variables based on the presence (Yes) or absence (No) of diarrhea, fever, and pneumonia(cough) frequency within the two weeks during baseline and end-line data collection. This may be categorize participants based on the response given.

CONTACTS AND LOCATIONS:
Overall Officials: Tadele Amente, Principal Investigator — Jimma University
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
Based on the progress of the study, I will decide to plan for future